CLINICAL TRIAL: NCT03962465
Title: Phase I Study of Inotuzumab Ozogamicin With 3 and 4 Drug Augmented Berlin-Frankfurt-Münster (BFM) Re-Induction for Patients With Relapsed or Refractory B-cell Acute Lymphoblastic Leukemia (B-ALL)
Brief Title: Phase I Study of Inotuzumab With Augmented BFM Re-Induction for Patients With Relapsed/Refractory B-cell ALL
Acronym: ALL-001
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Pfizer (Industry); Vanderbilt University (Other); University of Wisconsin, Madison (Other); Virginia Commonwealth University (Other)
Responsible Party: Principal Investigator, Michael Douvas, MD, Associate Professor of Medicine and Pediatrics, University of Virginia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21417
Record Dates: First submitted 2019-05-22; First posted 2019-05-24 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma | interventions — Inotuzumab Ozogamicin; Prednisone; Daunorubicin; Vincristine; Cytarabine; Methotrexate; pegaspargase

STUDY DESIGN:
Intervention Model Description: This is an early-phase study evaluating the safety of inotuzumab ozogamicin administered in combination with a 3-drug and 4-drug re-induction regimen in participants with relapsed or refractory B-ALL. The trial is planned to first determine the maximum tolerated dose (MTD) of the 3-drug re-induction regimen in Part 1 and then to determine the MTD of the 4-drug re-induction regimen (including pegaspargase) in Part 2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 3-drug re-induction regimen with inotuzumab (Experimental): One cycle of a 3-drug regimen comprised of standard doses of prednisone, vincristine, and daunorubicin with inotuzumab ozogamicin at a reduced dose.
  Intrathecal methotrexate (IT-methotrexate) and intrathecal cytarabine (IT-Ara-C) will be included for CNS prophylaxis.
  IV inotuzumab ozogamicin will be given at a reduced dose (may vary from a total cycle dose of 0.4 mg/m^2 to 0.9 mg/m^2)
  Interventions: Drug: Inotuzumab ozogamicin; Drug: Prednisone Pill; Drug: Daunorubicin; Drug: Vincristine; Drug: Cytarabine; Drug: Methotrexate
- 4-drug re-induction regimen with inotuzumab (Experimental): One cycle of a 4-drug regimen comprised of standard doses of prednisone, vincristine, daunorubicin, and pegaspargase with inotuzumab ozogamicin at a reduced dose.
  Intrathecal methotrexate (IT-methotrexate) and intrathecal cytarabine (IT-Ara-C) will be included for CNS prophylaxis.
  IV inotuzumab ozogamicin will be given at a reduced dose (may vary from a total cycle dose of 0.4 mg/m^2 to 0.9 mg/m^2)
  Interventions: Drug: Inotuzumab ozogamicin; Drug: Prednisone Pill; Drug: Daunorubicin; Drug: Vincristine; Drug: Cytarabine; Drug: Methotrexate; Drug: Pegaspargase

INTERVENTIONS:
Drug: Inotuzumab ozogamicin — By IV, given on days 12 and 19 Inotuzumab ozogamicin is approved as a single-agent in this population (patients with B-ALL) but adding it to these drug combinations has not been tested in humans
  Other Names: Besponsa
Drug: Prednisone Pill — Taken daily days 1-28 by mouth
  Other Names: Deltasone
Drug: Daunorubicin — By IV, given on days 1, 8, 15, and 22
  Other Names: Cerubidine; daunomycin; rubidomycin
Drug: Vincristine — By IV, given on days 1, 8, 15, and 22
  Other Names: Oncovin; Vincasar; Leurocristine
Drug: Cytarabine — Intrathecal, administered on day 1 only
  Other Names: Ara-C; Cytosar-U
Drug: Methotrexate — Intrathecal, administered on days 8 and 29
  Other Names: Otrexup; Rasuvo; Rheumatrex; Trexall; MTX; Amethopterin
Drug: Pegaspargase — By IV, given on day 4
  Other Names: Oncospar
  Arms: 4-drug re-induction regimen with inotuzumab

SUMMARY:
In the proposed study, escalating doses of inotuzumab ozogamicin will be added to a standard pediatric inspired re-induction regimen and administered to patients with relapsed or refractory B-cell acute lymphoblastic leukemia (B-ALL). Two re-induction regimens will be tested (one without pegaspargase and one including pegaspargase) and participants will be followed for disease status, allogeneic hematopoietic cell transplant (allo HCT), veno-occlusive disease following allo HCT, and overall survival.

DETAILED DESCRIPTION:
Inotuzumab ozogamicin has been studied as a single agent in refractory and relapsed ALL. In the relapsed setting, inotuzumab ozogamicin has been shown to achieve complete remission (CR) in 81% of patients and minimal residual disease (MRD) negativity in 78% of patients who achieve CR. In the proposed study, escalating doses of inotuzumab ozogamicin will be added to a standard pediatric inspired re-induction regimen and administered to patients with relapsed or refractory B-cell ALL. Two re-induction regimens will be tested. The first regimen is a 3-drug regimen comprised of prednisone, vincristine, and daunorubicin. The second is a 4-drug regimen comprised of prednisone, vincristine, daunorubicin, and pegaspargase. Intrathecal methotrexate (IT-methotrexate) and intrathecal cytarabine (IT-ARA-C) will be included for central nervous system (CNS) prophylaxis with both the 3-drug and 4-drug regimens. We hypothesize that combining inotuzumab ozogamicin with these regimens is safe and will improve CR rates, successful transition to allo HCT, and overall survival in patients with relapsed or refractory B-ALL.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Diagnosed with CD-22 positive* B-cell Acute Lymphoblastic Leukemia or B-cell Lymphoblastic Lymphoma (Philadelphia chromosome negative) * For the purposes of this study, CD-22 positive will be defined based on the analysis completed for diagnostic purposes.
4. Male or female, aged 16-60 years
5. ECOG performance status of 0-2
6. Left ventricular ejection fraction ≥ 50% measured by echocardiogram or MUGA
7. Either relapsed following remission after initial induction therapy or refractory to induction therapy
8. Adequate organ function, including serum creatinine ≤ 1.6 mg/dL OR creatinine clearance >50 ml/min by Cockgroft-Gault formula, bilirubin ≤ 1.5 mg/dL (except in patients with Gilbert's disease), AST, ALT and alkaline phosphatase ≤ 3 x upper limit of normal (elevation exceeding this threshold of either AST OR ALT would not meet eligibility)
9. For females of reproductive potential: negative pregnancy test
10. For females and males of reproductive potential: agreement to use adequate contraception during study participation and for an additional 1 year after the end of study treatment
11. Agreement to adhere to Lifestyle Considerations throughout study duration and for 1 year following last study treatment.

Exclusion Criteria:

1. Past receipt of a total of ≥ 300 mg/m^2 doxorubicin equivalents (600 mg/m^2 daunorubicin, 60 mg/m^2 idarubicin, 75 mg/m^2 mitoxantrone)
2. Current or past history of pancreatitis
3. QT interval on electrocardiogram (ECG) > 0.45 by Framingham formula
4. Known congestive heart failure
5. Known allergy to asparaginase (only an exclusion criteria for participants enrolling in part 2)
6. Presence of central nervous system (CNS) disease
7. Pregnancy or lactation
8. Chronic liver disease including chronic active hepatitis and/or cirrhosis
9. Active Hepatitis B virus (HBV) by core antibody, surface antigen (HBsAg) or viral load
10. Active Hepatitis C virus (HCV) (positive antibody test confirmed by viral load if antibody test is positive)
11. Known history of infection with Human Immunodeficiency Virus (HIV)
12. Active or uncontrolled infections
13. Abnormal baseline hepatic ultrasound (including Dopplers)
14. Prior allogeneic stem cell transplant
15. Prior use of inotuzumab ozogamicin
16. Known diagnosis of hemochromatosis with iron overload
17. Treatment with steroids or hydroxyurea for more than 7 days with each within the 2 weeks prior to registration -that is, each is allowed for up to 7 days
18. Gastrointestinal tract disease causing the inability to take oral medication, malabsorption syndrome, a requirement for intravenous (IV) alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease, or inability to swallow medications.
19. Philadelphia chromosome positive B-cell ALL

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-07-22 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Characterization of Adverse Events (CTCAE version 5) | All adverse events occurring through 30 days following last dose of inotuzumab ozogamicin.
  A characterization of all adverse events experienced by patients receiving these drug combinations. Also, any SAEs deemed related to study treatment, including veno-occlusive disease, will be captured at any time while the participant is on-study.
Dose-limiting toxicities | From initiation of inotuzumab ozogamicin through 30 days following the last dose of inotuzumab ozogamicin
  The number of dose-limiting toxicities will be used to determine the maximum tolerated dose combination for these combinations of drugs
Informative course of treatment | For each participant, up to the 29 days of study treatment
  Percent of patients that receive enough treatment to be informative to the study

CONTACTS AND LOCATIONS:
Overall Officials: Michael Douvas, MD, Principal Investigator — University of Virginia
Locations (4):
- United States (4):
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Virginia, Charlottesville, Virginia
  - VCU Massey Cancer Center, Richmond, Virginia
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No